CLINICAL TRIAL: NCT01658345
Title: Prognostic Importance of Microvascular Dysfunction in Asymptomatic Patients With Aortic Stenosis (PRIMID-AS)
Brief Title: Microvascular Dysfunction in Aortic Stenosis
Acronym: PRIMID-AS
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 87768
Record Dates: First submitted 2012-07-06; First posted 2012-08-07 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Aortic Stenosis
Keywords: aortic stenosis; asymptomatic; microvascular dysfunction; Cardiac MRI
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — With consent, a blood sample (up to 50ml) will be drawn and banked for prospective research studies. All research projects will be related to cardiovascular disease and approved by the Trial Steering Committee (TSC) or a committee delegated this responsibility by the TSC.
  All tissue will be collected, stored and disposed of in accordance with the Codes of Practice as laid out by the Human Tissue Authority.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aortic stenosis (AS), or narrowing of the aortic valve, is the commonest condition requiring valve surgery in the developed world. It is currently not known what determines who will go on to develop symptoms. Exercise testing may be able to identify these patients better than the severity of the narrowing itself, but with some limitations.

The purpose of this study is to compare whether MRI scanning or exercise testing can better identify patients with AS who are likely to benefit from surgery.

Design: The investigators will measure blood flow to the heart muscle with MRI scanning and perform exercise testing in 170 patients with AS and follow them for up to up to 2 years. Expected outcomes: MRI scanning will more accurately identify those patients with AS who will need surgery during this period. Anticipated Health Benefits: improved selection of patients with AS who are likely to benefit from early surgery. This is likely to reduce deaths in such patients.

DETAILED DESCRIPTION:
Surgical AVR remains the universally accepted management for symptomatic aortic stenosis (AS). However, the best management of severe aortic stenosis, in the absence of symptoms, remains one of the most controversial areas in modern Cardiology.

Exercise testing can identify asymptomatic patients with AS at increased risk, but with limited specificity. In a BHF funded project, the investigators have identified that cardiac MRI measured Myocardial Perfusion Reserve (MPR) may be a novel imaging biomarker in AS. MPR was the only independent predictor of aerobic exercise capacity (peak VO2) in patients with severe AS and was also inversely related to symptomatic status.

In this multi-centre, observational, cohort outcome study, the investigators will follow 175 patients with asymptomatic moderate to severe AS for a minimum of 12 months, and determine whether MPR is a better predictor of outcome than exercise testing, elucidate the mechanisms contributing to symptom development in AS and establish the determinants of MPR in AS. Patients will be recruited from tertiary Cardiac centres, as well as regional hospitals. Comprehensive CMR with adenosine stress to determine LV mass and function, focal and diffuse fibrosis and MPR; cardiopulmonary exercise testing (peak VO2 and exercise symptoms); rest and exercise echocardiography (AS severity, valve compliance) and NT-proBNP will be performed. The study will be run in conjunction with the Glasgow CTU. Investigations will be analysed blind to patient status and data will be entered in a validated database. Statistical analysis will be performed under the supervision of Prof. Ian Ford. The relationship between MPR and exercise testing with 1-year outcome will be analysed using logistic regression. Paired comparisons of the specificities of the two approaches on the same dataset will be carried out using McNemar's test.

The primary hypothesis is that MPR will be a better predictor of adverse outcome than exercise testing.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate-severe aortic stenosis (2 or more of: AVA < 1.5cm2, peak PG >36mmHg or mean PG > 25mmHg).
2. Asymptomatic.
3. Age > 18 years and < 85 years.
4. Prepared to consider AVR if symptoms develop.
5. Ability to perform bicycle exercise test

Exclusion Criteria:

1. History of CABG or MI within previous 6 months.
2. Severe valvular disease other than AS.
3. Previous Valve surgery
4. Persistent Atrial Fibrillation or Flutter
5. History of Heart Failure
6. Severe Asthma.
7. Severe renal impairment eGFR < 30ml/min.
8. Planned aortic valve replacement.
9. Significant LV systolic dysfunction (EF < 40%)
10. Any absolute contraindication to CMR
11. Any absolute contraindication to Adenosine
12. Participation in an Interventional Clinical Trial at Inclusion.
13. Other medical condition that limits life expectancy or precludes AVR.
14. Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiology outpatients department and echocardiography department.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Typical AS Symptoms necessitating AVR. | 12 months
Cardiovascular death. | 12 months
Major adverse cardiovascular events (MACE) | 12 months
  MACE: hospitalisation with heart failure, chest pain, syncope, arrhythmia or stroke

SECONDARY OUTCOMES:
Individual components of primary composite outcome measures. | Upto 2 years.
  Typical symptoms requiring referral for AVR, cardiovascular death, Major adverse cardiovascular events.
Development of typical symptoms, AVR, death from any cause or MACE during the entire study period. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gerry P McCann, MBChB, MD, Principal Investigator — University of Leicester
Locations (3):
- United Kingdom (3):
  - Glenfield Hospital, Leicester, Leicestershire
  - Leeds General Infirmary, Leeds, West Yorkshire
  - University of Glasgow, Glasgow

REFERENCES:
- [Background] Steadman CD, Jerosch-Herold M, Grundy B, Rafelt S, Ng LL, Squire IB, Samani NJ, McCann GP. Determinants and functional significance of myocardial perfusion reserve in severe aortic stenosis. JACC Cardiovasc Imaging. 2012 Feb;5(2):182-9. doi: 10.1016/j.jcmg.2011.09.022. PMID 22340825
- [Background] McCann GP, Steadman CD, Ray SG, Newby DE; British Heart Valve Society. Managing the asymptomatic patient with severe aortic stenosis: randomised controlled trials of early surgery are overdue. Heart. 2011 Jul;97(14):1119-21. doi: 10.1136/hrt.2011.223800. Epub 2011 Mar 12. No abstract available. PMID 21398695
- [Background] Steadman CD, Ray S, Ng LL, McCann GP. Natriuretic peptides in common valvular heart disease. J Am Coll Cardiol. 2010 May 11;55(19):2034-48. doi: 10.1016/j.jacc.2010.02.021. PMID 20447526
- [Background] Das P, Rimington H, Chambers J. Exercise testing to stratify risk in aortic stenosis. Eur Heart J. 2005 Jul;26(13):1309-13. doi: 10.1093/eurheartj/ehi250. Epub 2005 Apr 8. PMID 15820999
- [Derived] Chan DCS, Singh A, Greenwood JP, Dawson DK, Lang CC, Berry C, Pakkal M, Everett RJ, Dweck MR, Ng LL, McCann GP. Effect of the 2017 European Guidelines on Reclassification of Severe Aortic Stenosis and Its Influence on Management Decisions for Initially Asymptomatic Aortic Stenosis. Circ Cardiovasc Imaging. 2020 Dec;13(12):e011763. doi: 10.1161/CIRCIMAGING.120.011763. Epub 2020 Dec 8. PMID 33287584
- [Derived] Graham-Brown MP, Singh AS, Gulsin GS, Levelt E, Arnold JA, Stensel DJ, Burton JO, McCann GP. Defining myocardial fibrosis in haemodialysis patients with non-contrast cardiac magnetic resonance. BMC Cardiovasc Disord. 2018 Jul 13;18(1):145. doi: 10.1186/s12872-018-0885-2. PMID 30005636
- [Derived] Singh A, Greenwood JP, Berry C, Dawson DK, Hogrefe K, Kelly DJ, Dhakshinamurthy V, Lang CC, Khoo JP, Sprigings D, Steeds RP, Jerosch-Herold M, Neubauer S, Prendergast B, Williams B, Zhang R, Hudson I, Squire IB, Ford I, Samani NJ, McCann GP. Comparison of exercise testing and CMR measured myocardial perfusion reserve for predicting outcome in asymptomatic aortic stenosis: the PRognostic Importance of MIcrovascular Dysfunction in Aortic Stenosis (PRIMID AS) Study. Eur Heart J. 2017 Apr 21;38(16):1222-1229. doi: 10.1093/eurheartj/ehx001. PMID 28204448
- [Derived] Singh A, Ford I, Greenwood JP, Khan JN, Uddin A, Berry C, Neubauer S, Prendergast B, Jerosch-Herold M, Williams B, Samani NJ, McCann GP. Rationale and design of the PRognostic Importance of MIcrovascular Dysfunction in asymptomatic patients with Aortic Stenosis (PRIMID-AS): a multicentre observational study with blinded investigations. BMJ Open. 2013 Dec 18;3(12):e004348. doi: 10.1136/bmjopen-2013-004348. PMID 24353258